CLINICAL TRIAL: NCT04894578
Title: Can Reverse Oblique Distal Minimal-invasive Osteotomies Replace Arthrodesis of the Tarsometatarsal Joints? - a Prospective, Comparative Trial of 50 Patients
Brief Title: A Comparative Trial of a Minimal-invasive Technique Versus Open Arthrodesis in the Treatment of Midfoot Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kantonsspital Baden (Other)
Responsible Party: Principal Investigator, Christopher G Lenz, Principal Investigator, Kantonsspital Baden
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-00916
Record Dates: First submitted 2021-05-11; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Osteoarthritis; Foot; Osteotomy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Patients suffering from midfoot arthritis after failed prior conservative therapy who undergo a reverse distal metatarsal minimal-invasive osteotomy
  Interventions: Procedure: reverse distal metatarsal minimal-invasive osteotomy
- Group B (Active Comparator): Patients suffering from midfoot arthritis after failed prior conservative therapy who undergo a fusion of one or more midfoot (tarsometatarsal) joints
  Interventions: Procedure: tarsometatarsal fusion

INTERVENTIONS:
Procedure: reverse distal metatarsal minimal-invasive osteotomy — minimal-invasive oblique osteotomy of the two or three metatarsal bones using a straight burr
  Arms: Group A
Procedure: tarsometatarsal fusion — open procedure with fusion and screw and plate fixation of two to three tarsometatarsal joints
  Arms: Group B

SUMMARY:
Group A: Patients suffering from midfoot arthritis after failed prior conservative therapy who undergo a reverse distal metatarsal minimal-invasive osteotomy Group B: Patients suffering from midfoot arthritis after failed prior conservative therapy who undergo a fusion of one or more midfoot (tarsometatarsal) joints

DETAILED DESCRIPTION:
Midfoot arthritis is a common condition leading to disabling chronic foot pain that affects activities of daily living. The causes can be primary osteoarthritis (OA), inflammatory or post-traumatic. We are looking at OA of the lesser (second and/or third) tarsometatarasal joints (TMTJ). Orthotics, customised shoes or steroid injections are options to treat this condition nonoperatively. If these measures fail, arthrodesis of the arthritic joints represents the standard procedure to surgical treatment. Generally, the results of this procedure are at a satisfactory level for the patients, nevertheless, there is a relevant amount of patients with residual pain, lack of a normal foot appearance, and the need for unplanned surgery or use of orthotics postoperatively. Furthermore, patients undergoing an arthrodesis of the lesser TMTJ usually have to stay in hospital for 4-7 days. Postoperatively, patients are only allowed to partially weightbear for at least 6 weeks and need a cast for six weeks as well. During that time thrombosis prophylaxis is administered for about 6 weeks.

The conventional distal minimal-invasive metatarsal osteotomy (DMMO) is an accepted technique for metatarsal osteotomies. Recently, Schneider et al. presented results of a modification of the conventional DMMO, the reverse DMMO to treat OA of the lesser TMTJ, thus representing an alternative treatment to arthrodesis. The procedure has many benefits. It allows outpatient care, an immobilisation in a cast is not necessary. Instead, patients have to wear a flat postoperative shoe for 2-3 weeks and are allowed to fully weightbear from day one after surgery. Therefore, thrombosis prophylaxis is not necessary unless there are specific risk factors.

However, while the arthrodesis directly addresses the arthritic joints, the R-DMMO alters the ground reaction force of the metatarsal head leading to less stress at the level of the TMTJ, but the arthritic joint itself is not approached. Still, the results presented by Schneider et al. are promising. Since there was no group to compare the treatment with, the small sample size, and a retrospective design, we would like to prospectively compare these two surgical procedures directly in order to find out whether or not the R-DMMO can be recommended as a standard procedure for OA of the lesser TMTJ at a much more convenient level for patients regarding the whole perioperative protocol. No vulnerable population is included. The scientific value is remarkable since this would be the first study to examine this matter and we are able to provide a high level of evidence due to the prospective-randomised and comparative design of the study. All legal requirements will be fulfilled and the ethical standards are guaranteed.

Both procedures have been described and the technique of the DMMO itself is not new, but its modification (R-DMMO) represents a new approach for this condition. Both procedures are reliable and safe, which is why the risk category of the study is A according to ClinO, Art. 61.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Midfoot arthritis of lesser TMTJ (second, third, rarely fourth and fifth) with ongoing disabling pain
* Able to give informed consent as documented by signature
* failed conservative treatment for a period of at least 3 months (CSI injections and/or orthotic devices)

Exclusion Criteria:

* Concomitant fusion of 1st TMTJ
* Patients younger than 18 years
* Contraindication to undergo surgery or general anaesthesia
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-14 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcome using a patient related outcome measure, the FAAM score (Validated Foot and Ankle Ability Measure). The score is a self-report outcome instrument developed to assess physical function. The change between the time points is measured. | 6 weeks, 3 months, 6 months, 12 and 24 months post surgery
  FAAM score, the highest score is 100, indicating the best possible outcome

SECONDARY OUTCOMES:
Duration of procedure | through study completion, an average of 2 years
  Duration of procedure (in minutes from first incision until wound is closed)
Length of hospital stay | through study completion, an average of 2 years
  Length of hospital stay in days
Visual Analogue Scale (VAS) score. It is a measurement instrument for the amount of pain that a patient feels. The score is assessed preoperatively and the change between the time points is measured. | 6 weeks, 3 months, 6 months, 12 and 24 months post surgery
  Pain score (scale 0-10, where 10 is the maximum pain)
Radiological union by evaluating conventional X-Ray. Preoperative X-Rays and postoperative X-Rays are comparted and the change in union in terms of bone densitiy is assessed postoperatively. | 6 weeks, 3 months, 6 months, 12 and 24 months post surgery
  Union of bone on conventional X-Ray in two planes (dorsoplantar and lateral views)
Complications | 6 weeks, 3 months, 6 months, 12 and 24 months post surgery
  Identifying minor and major complications of the procedure (e.g. infections)

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Baden, Baden, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gougoulias N, Lampridis V. Midfoot arthrodesis. Foot Ankle Surg. 2016 Mar;22(1):17-25. doi: 10.1016/j.fas.2015.04.004. Epub 2015 Apr 24. PMID 26869495
- [Background] Laffenetre O, Perera A. Distal Minimally Invasive Metatarsal Osteotomy ("DMMO" Procedure). Foot Ankle Clin. 2019 Dec;24(4):615-625. doi: 10.1016/j.fcl.2019.08.011. PMID 31653366
- [Background] Schneider TE, Varrall CR, Malhotra K. Early results of minimally invasive, reverse-oblique, distal metaphyseal metatarsal osteotomy (R-DMMO) for arthritis of the lesser tarsometatarsal joints - A retrospective case series. Foot (Edinb). 2020 Jun;43:101652. doi: 10.1016/j.foot.2019.10.007. Epub 2019 Oct 25. PMID 32086136